CLINICAL TRIAL: NCT06822634
Title: Advances in Imaging to Assess Response in Rectal Cancer (AIR-REC)
Brief Title: Advances in Imaging to Assess Response in Rectal Cancer
Acronym: AIR-REC
Status: Recruiting | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: GN23ON218; 329328 (Other: IRAS)
Record Dates: First submitted 2025-01-14; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer (CRC)
Keywords: Colorectal cancer; colorectal cancer (crc); CRC; MRI
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample, biopsy sample and stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Colorectal cancer patients: Patients with histologically confirmed invasive rectal adenocarcinoma
  Interventions: Other: Observational single centre feasibility study

INTERVENTIONS:
Other: Observational single centre feasibility study — Patients scheduled to undergo standard of care neo. adjuvant radiotherapy prior to surgery.

SUMMARY:
The goal of this observational study is to determine the feasibility of acquiring serial MRI images for advanced radiotherapy planning in colorectal patients.

The main question it aims to answer:

Is it feasible to acquire serial MR images for advanced radiotherapy planning for rectal cancer.

DETAILED DESCRIPTION:
Bowel cancer is the 4th most common cancer in the UK and accounts for 11% of all new cancer diagnoses, a third of these cancers are located in the rectum. Approximately 732, 000 rectal cancers are diagnosed in Europe per year.

Radiotherapy (RT) is a well-established treatment for locally advanced rectal cancer (LARC). It can be used pre operatively in margin threatening disease to increase the likelihood of R0 resection margins; reduce the rate of loco regional recurrence; and to improve loco regional control for patients unsuitable for surgery. There are two treatment regimes used internationally, with strong evidence from numerous randomised clinical trials. These are long course chemoradiotherpy (LCRT) with a dose of 45-60Gy delivered in 25 fractions and short course radiotherapy (SCRT) with a dose of 25Gy in 5 fractions. No long-term superiority of either approach has been found thus far.

RT indications for LARC are defined by clinic-radiological MRI defined criteria. Accurate and precise delineation of the target volume is fundamental to the success of RT. CT planning scans are traditionally used for target delineation in RT, have poor soft tissue contrast and on this dataset have shown overestimation of tumour volumes. Given that magnetic resonance images (MRI) brings superior visualisation of soft tissue in the diagnostic phase of LARC, there has been a move towards routine use of MRI within the delivery of RT.

MRI imaging is considered the gold standard in the staging and response assessment of rectal cancers. The rectum lends well to the exquisite soft tissue definition MRI offers, and additional functional information can be used to further characterise tumour. Improved tumour localisation up front and assessment of responses during RT has the potential to improve patient outcomes in numerous ways.

The use of MRI in RT planning of rectal cancer is relatively new. A survey of UK practice identified specifically 64% of centres use a diagnostic MRI alongside to aid delineation, 28% register MRI images with the diagnostic scan and only 3% use a registered scan in the RT position. National rectal cancer guidelines recommend MRI to be used if possible to aid delineation of the gross tumour volume (GTV). A report published by IPEM gives clear guidance for the optimal use in RT planning for rectal cancer.

There is a general acceptance that the use of MRI in rectal cancer RT planning is superior. In the literature there are a number of studies looking at different aspects of MRI application in the rectal cancer RT pathway. However, there is great disparity in the focus of these research papers.

One of the main challenges in gaining optimal benefit from this technology is the many uncertainties in the planning and delivery of RT to rectal cancers. Largely due to the target being a soft tissue structure, which moves independently due to gas and faecal filling. The surrounding elective volume includes the mesorectum and regional lymph nodes, resulting in targets with a differential motion. This brings more uncertainty in reproducibility, the foundation of accurate and precise RT. MRI with improved soft tissue visualisation could potentially enable voluming of only the tumour and not the full rectal lumen. This could be practice changing and requires careful consideration in implementation. For these reasons correct application of MRI in rectal cancer RT planning is crucial to ensure the optimal benefit from this technology is gained. In the setting of serial imaging reproducibility is more important, where repeatability and reliability of data matters more.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed rectal adenocarcinoma.
* T stage 3b or above and/or high risk factors eg. EMVI, nodal disease.
* Participant able to give written informed consent.
* Male or non-pregnant female ≥18 years of age.
* Scheduled to undergo radical radiotherapy.
* Patients willing and able to comply with the protocol for the duration of study.

Exclusion Criteria:

* Contra-indications to MRI, such as claustrophobia, excessive body weight, MRI unsafe implants, ferrous metal in the body, insufficient information on prior surgeries. MRI conditional implants where conditions cannot be met (e.g pacemakers).
* Any previous radiotherapy to the pelvis.
* Inflammatory bowel disease.
* Other severe or uncontrolled systemic disease or evidence of any other significant disorder or lab finding that makes it undesirable for the patient to participate in the study, as determined by the treating clinician.
* History of physical or psychiatric disorder that would prevent informed consent and compliance with the protocol.
* Patients with de-functioning stoma.
* Major surgery within 28 days prior to trial entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be locally advanced rectal cancer patients with histologically confirmed rectal adenocarcinoma.
  20 patients will be recruited to the study.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-06-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Feasibility of acquiring serial MRI for advanced radiotherapy planning of rectal cancer. | 18 months
  Feasibility defined as 70% of study participants completing a baseline and repeat scan acquisition.

SECONDARY OUTCOMES:
Volumetric radiotherapy target volume data- longitudinal changes in radiotherapy target volume data measured in cubic centimetres | 18 Months
  Identify anatomical changes in radiotherapy target volume from baseline and repeat scans measured in cubic centimetres.
Quantification of MR image parameters- extraction of apparent diffusion coefficient (ADC) from defined radiotherapy target volumes on functional MR images | 18 months
  Feasibility of measuring apparent diffusion coefficient (ADC) using functional MR sequences on baseline and repeat scans, defined as a quantified value in mm²/s (square millimetres per second).
Quantify inter-observer target delineations | 18 months
  Quantify inter-observer variation in target delineations on CT and MRI sequences.
  Record inter observer agreement metrics and volume between observers on CT and MRI datasets.
Health-related quality of life of study participant using European Organisation for Research and Treatment of Cancer patients' validated tools EORTC QLQ CR30 and EORTC CR 29 | 18 months
  To measure health related quality of life of study participants validated tools EORTC QLQ CR30 and EORTC CR 29.

CONTACTS AND LOCATIONS:
Overall Officials: Ms Lynsey Devlin, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Beatson West of Scotland Cancer Centre, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Currently undecided